CLINICAL TRIAL: NCT01023100
Title: A Study In Trained Taste Panel Healthy Adult Volunteers To Investigate The Palatability Of Select Formulations Of CP-690,550 Oral Solution
Brief Title: A Study Of The Taste Of Different Oral Liquid Preparations Of CP-690,550 In Trained Adult Product Testers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A3921115
Record Dates: First submitted 2009-11-25; First posted 2009-12-02 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: taste study open label investigational drug oral therapy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental)
  Interventions: Drug: CP 690,550 oral solutions

INTERVENTIONS:
Drug: CP 690,550 oral solutions — flavored and unflavored prototype CP-690,550 formulations

SUMMARY:
This study will test the palatability of several different CP-690,550 oral preparations in trained product tester healthy volunteers.

DETAILED DESCRIPTION:
To develop a palatable pediatric oral solution dosage form of CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Trained healthy non-pregnant product testers, age 18-75

Exclusion Criteria:

* Severe acute or chronic medical conditions, including hepatitis or tuberculosis infections or clinically significant laboratory abnormalities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
A complete description of the sensory attributes of products (eg, aroma, flavor, texture, and mouthfeel). | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Woburn, Massachusetts, United States